CLINICAL TRIAL: NCT02195921
Title: Acupuncture for Chemotherapy-Induced Nausea and Vomiting: A Randomized Clinical Trial
Brief Title: Acupuncture for Chemotherapy-Induced Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yi Guo, Dean of Traditional Chinese Medicine School, Tianjin University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014CB543201-02
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Single point CV12 (Experimental): choose single point:Zhongwan(CV12).Zhongwan(CV12):On the upper abdomen, 4 B-cun superior to the centre of the umbilicus, on the anterior median line.Manipulating until achieving a "de Qi" sensation,then the needle is connected through a electro-acupuncture apparatus,the positive pole is linked to the needle, and the reference pole is located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA.The operation lasts for 30 min. The treatmeat is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days. Received routine antiemetic treatment.
  Interventions: Other: single point Zhongwan(CV12) plus antiemetic drug
- Single point ST36 (Experimental): choose another single point Zusanli（ST36）.Zusanli(ST36):On the anterior aspect of the leg, on the line connecting ST35 with ST41, 3 B-cun inferior to ST35，located on the tibialis anterior muscle..Manipulating until achieving a "de Qi" sensation, then the needle is connected through a electro-acupuncture apparatus,the positive pole is linked to the needle, and the reference pole is located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA.The operation lasts for 30 min. The treatmeat is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days. Received routine antiemetic treatment.
  Interventions: Other: single point Zusanli(ST36) plus antiemetic drug
- ST36+CV12 acupoints (Experimental): Choose both Zusanli(ST36) and Zhongwan（CV12）.Manipulating until achieving a "de Qi" sensation, then the needle is connected through a electro-acupuncture apparatus,the positive pole is linked to the needle, and the reference pole is located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA.The operation lasts for 30 min. The treatmeat is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days. Received routine antiemetic treatment.
  Interventions: Other: Zusanli(ST36)and Zhongwan(CV12) plus antiemetic drug
- only antiemetics (Active Comparator): The control group will receive standard antiemetics alone. Standard antiemetics for all groups are based on American Society of Clinical Oncology clinical practice guideline. 5-hydroxytryptamine-3 (5-HT3) antagonist (Ramosetron , Tropisetron)and dexamethasone are supplied from the first day of chemtherapy,and lasting for 3-5days. If nausea and/or vomiting is persistent and failed to respond to the antiemetic treatment , based on the experience of each clinician, the other advanced 5-HT3 antagonist or a neurokinin 1 antagonist(NK-1) will be chosen.
  Interventions: Drug: only antiemetic drug

INTERVENTIONS:
Other: single point Zhongwan(CV12) plus antiemetic drug — All participants were supine in the hospital bed. A disposable sterile acupuncture needle (ø 0.30 × 40 mm, Hwato) was inserted vertically at approximately 20-30 mm until "De Qi" (sensation of soreness, numbness, distension, etc. around the acupoint) was reported by the participants. Then, the needle handle was clamped via a metal clip to connect to the positive electrode of the electric acupuncture apparatus (Huatuo, SDZ-V model, Suzhou Medical Appliance). Another reference electrode was placed 1 cm above the CV12 acupoints of the stimulation point, where no acupoints or meridians passed through. A dilatational wave at a frequency of 2/10 Hz and a current intensity at the highest level tolerated by the patient, with a maximum intensity no more than 10 mA, were used to deliver the EA stimulation. People in the intervention groups were offered a standardized 30-minute EA session once daily from the 1st day of the four-day chemotherapy cycle.
  Arms: Single point CV12
Other: single point Zusanli(ST36) plus antiemetic drug — A disposable sterile acupuncture needle (ø 0.30 × 40 mm, Hwato) was inserted vertically at approximately 20-30 mm until "De Qi" (sensation of soreness, numbness, distension, etc. around the acupoint) was reported by the participants. Then, the needle handle was clamped via a metal clip to connect to the positive electrode of the electric acupuncture apparatus (Huatuo, SDZ-V model, Suzhou Medical Appliance). Another reference electrode was placed 1cm below ST36 acupoints of the stimulation point, respectively, where no acupoints or meridians passed through. A dilatational wave at a frequency of 2/10 Hz and a current intensity at the highest level tolerated by the patient, with a maximum intensity no more than 10 mA, were used to deliver the EA stimulation. People in the intervention groups were offered a standardized 30-minute EA session once daily from the 1st day of the four-day chemotherapy cycle.
  Arms: Single point ST36
Other: Zusanli(ST36)and Zhongwan(CV12) plus antiemetic drug — Stimulating both Zusanli(ST36)and Zhongwan(CV12)
  Arms: ST36+CV12 acupoints
Drug: only antiemetic drug — received routine antiemetic treatment
  Arms: only antiemetics

SUMMARY:
The purpose of this study is to clarify whether the matching acupoints is more effective than a single point by electroacupuncture in the management of chemotherapy-induced nausea and vomiting .

DETAILED DESCRIPTION:
Patients were assigned to Four sessions of electroacupuncture(EA) at the CV12, ST36, CV12+ST36 acupoints or antiemetic therapy over 5 days. primary and secondary outcomes and Adverse Eventswill be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed as cancer and need to accept chemotherapy.
2. The score of Karnofsky ≥70
3. Patients of either gender and older than 18 years
4. Patients receiving chemotherapy both outpatients and inpatients
5. Patients receiving chemotherapy either he first or multiple cycle, but the patient will be taken in only one time
6. To receive chemotherapy containing cisplatin(DDP≥75mg/m2) or joint chemotherapy programmes of Anthracyclines(Adriamycin≥40mg/m2 or epirubicin≥60mg/m2)
7. Life expectancy≥ 6 months
8. Willing to participate in the study and be randomized into one of the four study groups.

Exclusion Criteria:

1. To receive radiotherapy and chemotherapy
2. Gastrointestinal tumors
3. Patients with serious liver disease or abnormal hepatorenal function (AST,ACT, and TBIL are 3 times more than normal, BUN and Cr are 2 times more than normal)
4. Presence of cardiac pacemaker
5. Active skin infection
6. Nausea and/or vomiting resulting from opioids or metabolic imbalance (electrolyte disturbances)
7. Patients unable to provide self-care or communication
8. Nausea and/or vomiting resulting from mechanical risk factors (i.e., intestinal obstruction)
9. Brain metastases
10. Women in pregnant and lactating period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Guo, Study Director — Tianjin University of Traditional Chinese Medicine
Locations (1):
- Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Chen B, Guo Y, Zhao X, Gao LL, Li B, Zhao TY, Zhang QW, Zou JX, Li MY, Guo YM, Guo Y, Pan XF. Efficacy differences of electroacupuncture with single acupoint or matching acupoints for chemotherapy-induced nausea and vomiting: study protocol for a randomized controlled trial. Trials. 2017 Oct 13;18(1):477. doi: 10.1186/s13063-017-2186-y. PMID 29029639

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 160 patients were enrolled randomly assigned to the CV12 (n = 40), ST36 (n = 40), DA (n = 40) and control (n = 40) groups. One participant in each of the CV12 and control groups was further excluded due to missing sessions, and one was excluded in the DA group because of repeated enrollment during the study period.
Groups:
- Single Point CV12: choose single point:Zhongwan(CV12).Zhongwan(CV12):On the upper abdomen, 4 B-cun superior to the centre of the umbilicus, on the anterior median line.Manipulating until achieving a "de Qi" sensation,then the needle is connected through a electro-acupuncture apparatus,the positive pole is linked to the needle, and the reference pole is located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA.The operation lasts for 30 min. The treatmeat is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days.
  single point Neiguan(CV12) plus antiemetic drug
- Single Point ST36: choose another single point Zusanli（ST36）.Zusanli(ST36):On the anterior aspect of the leg, on the line connecting ST35 with ST41, 3 B-cun inferior to ST35，located on the tibialis anterior muscle..Manipulating until achieving a "de Qi" sensation, then the needle is connected through a electro-acupuncture apparatus,the positive pole is linked to the needle, and the reference pole is located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA.The operation lasts for 30 min. The treatmeat is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days.
  single point Zusanli(ST36) plus antiemetic drug
- Matching Points ST36+CV12: Choose both Zusanli(ST36) and Zhongwan（CV12）.Manipulating until achieving a "de Qi" sensation, then the needle is connected through a electro-acupuncture apparatus,the positive pole is linked to the needle, and the reference pole is located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA.The operation lasts for 30 min. The treatmeat is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days.
  matching points Zusanli(ST36)and Neiguan(CV12) plus antiemetic drug
- Only Antiemetics: The control group will receive standard antiemetics alone. Standard antiemetics for all groups are based on American Society of Clinical Oncology clinical practice guideline. 5-hydroxytryptamine-3 (5-HT3) antagonist (Ramosetron , Tropisetron)and dexamethasone are supplied from the first day of chemtherapy,and lasting for 3-5days. If nausea and/or vomiting is persistent and failed to respond to the antiemetic treatment , based on the experience of each clinician, the other advanced 5-HT3 antagonist or a neurokinin 1 antagonist(NK-1) will be chosen.
  only antiemetic drug
Period: Overall Study
Arm/Group | Single Point CV12 | Single Point ST36 | Matching Points ST36+CV12 | Only Antiemetics
Started | 40 | 40 | 40 | 40
Completed | 39 | 39 | 39 | 40
Not Completed | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patient demographic characteristics were similar among the four groups at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Point CV12 | Single Point ST36 | Matching Points ST36+CV12 | Only Antiemetics | Total
Number analyzed (Participants) | 40 | 40 | 39 | 40 | 159
Age, Continuous [Median (Standard Deviation); unit: years] | 52 (7.23) | 55.4 (9.03) | 51.7 (11.37) | 53.7 (7.16) | 53 (8.954)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 30 | 29 | 114
  Male | 11 | 14 | 9 | 11 | 45
Region of Enrollment [Number; unit: participants]
  China | 40 | 40 | 39 | 40 | 159

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Nausea
Description: Percentage of participants with nausea was assessed by visual analog scale (VAS) ranging from 0 (no nausea) to 10 (worst nausea). A score of 0 means no nausea for a portion of the patient's assessment.
Time Frame: 5 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ST36+CV12: Choose both Zusanli(ST36) and Zhongwan（CV12）.Manipulating until achieving a "de Qi" sensation, then the needle is connected through a electro-acupuncture apparatus,the positive pole is linked to the needle, and the reference pole is located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA.The operation lasts for 30 min. The treatmeat is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days.
  matching points Zusanli(ST36)and Neiguan(CV12) plus antiemetic drug
Arm/Group | Single Point CV12 | Single Point ST36 | ST36+CV12 | Only Antiemetics
Number analyzed (Participants) | 39 | 39 | 39 | 40
percentage of participants | 31 [24 to 37] | 47 [40 to 54] | 54 [47 to 61] | 53 [46 to 60]

2. Primary Outcome: Number of Times Vomiting Occurs After Chemotherapy
Description: The number of times vomiting occurs after chemotherapy for each participant during 0-120 hours. The evaluator completed daily diaries for each time point.
Time Frame: 5 days
Measure: Mean (95% Confidence Interval); unit: number of times for patients
Groups:
- CV12: Stimulated CV12
- ST36: Stimulated ST36
- CV12+ST36: Stimulated CV12+ST36
- Control: Antiemetic only
Arm/Group | CV12 | ST36 | CV12+ST36 | Control
Number analyzed (Participants) | 39 | 39 | 39 | 40
number of times for patients | 0.44 [0.28 to 0.60] | 0.54 [0.35 to 0.74] | 0.78 [0.52 to 1.05] | 0.53 [0.32 to 0.74]

3. Primary Outcome: Rhodes Index of Nausea, Vomiting and Retching
Description: The RINVR scale has 8 items . The scale divides the occurrence of nausea , vomiting , and retching within 12 hours of tumor chemotherapy patients into 5 grades , which are scored from 0 to 4 points . The lower the score , the better . The RINVR scale can be divided into three dimensions : symptom experience time , symptom frequency and symptom severity .
Time Frame: 5 days
Population: Data were not collected.Due to its relatively weak specificity, the data was not collected. we replaced it with (visual analog scale) VAS and number of times of vomiting occurs which were recorded in the first and second primary outcome.
Arm/Group | CV12 | ST36 | CV12+ST36 | Control
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants With Nausea and Number of Times of Vomiting Occurs After Chemotherapy
Description: Rhodes Index of Nausea, Vomiting and Retching was replaced by percentage of participants with nausea (assessed by VAS) and number of times of vomiting occurs which were recorded in the first and second primary outcome.
Time Frame: 5 days
Reporting Status: Not Posted, anticipated posting 2020-12

5. Secondary Outcome: Grading of Constipation and Diarrhea
Description: The grading of constipation and diarrhea.We deleted this evaluation method due to weak correlation.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | Single Point CV12 | Single Point ST36 | Matching Points ST36+CV12 | Only Antiemetics
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Electrogastrogram
Description: We deleted this evaluation method due to weak correlation.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | Single Point CV12 | Single Point ST36 | Matching Points ST36+CV12 | Only Antiemetics
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: the Assessment of Quality of Life
Description: Assessed by the Functional Assessment of Cancer Treatment-General (FACT-G) .The FACT-G includes 27 items and is divided among 4 subscales: physical well-being (PWB), functional well-being (FWB), social/family well-being (SWB), and emotional well-being (EWB). The total FACT-G score ranges from 0 to 108 and is calculated by the sum of the subscales, with higher scores indicating greater functional status
Time Frame: 5 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Single Point CV12 | Single Point ST36 | Matching Points ST36+CV12 | Only Antiemetics
Number analyzed (Participants) | 39 | 39 | 39 | 40
score on a scale | 47 [43 to 50] | 47 [42.25 to 49] | 45 [36 to 47] | 45 [39 to 49]

8. Secondary Outcome: the Assessment of Anxiety and Depression
Description: Assessed by Hospital Anxiety and Depression Scale (HADS scale). It includes fourteen items, seven of which assess anxiety and the other seven assess depression (30). The total scores range from 0 to 21 for depression and anxiety, respectively, with higher scores indicating more depression and anxiety.
Time Frame: 5 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Single Point CV12 | Single Point ST36 | Matching Points ST36+CV12 | Only Antiemetics
Number analyzed (Participants) | 39 | 39 | 39 | 40
score on a scale | 8 [6 to 8] | 7 [6 to 8] | 8 [7 to 9] | 7 [6 to 9]

9. Other Pre Specified Outcome: Blood Routine Examination
Description: We deleted this evaluation method due to weak correlation.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | Single Point CV12 | Single Point ST36 | Matching Points ST36+CV12 | Only Antiemetics
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Other Pre Specified Outcome: Electrocardiogram
Description: We deleted this evaluation method due to weak correlation.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | Single Point CV12 | Single Point ST36 | Matching Points ST36+CV12 | Only Antiemetics
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Other Pre Specified Outcome: Hepatic and Renal Function
Description: We deleted this evaluation method due to weak correlation.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | Single Point CV12 | Single Point ST36 | Matching Points ST36+CV12 | Only Antiemetics
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Other Adverse Effect During the Chemotherapy
Time Frame: 5 days
Population: Recorded in Adverse Events
Arm/Group | Single Point CV12 | Single Point ST36 | Matching Points ST36+CV12 | Only Antiemetics
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 days after chemotherapy
Description: Electroacupuncture may be a safe treatment
Arm/Group | Single Point CV12 | Single Point ST36 | ST36+CV12 | Only Antiemetics
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 0/39 | 1/39 | 2/39 | 1/40
OTHER ADVERSE EVENTS (reported when occurring in more than 2.54% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Point CV12 (N=39) | Single Point ST36 (N=39) | ST36+CV12 (N=39) | Only Antiemetics (N=40)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No